CLINICAL TRIAL: NCT06308133
Title: Biological Variables Affecting CD34+ Peripheral Cells Collection Efficiency Using the Spectra Optia Continuous Mononuclear Cell Collection System: Hematocrit as Determinant for CD34+ Collection Efficency.
Brief Title: Biological Variables Affecting CD34+ Peripheral Cells Collection Efficiency
Acronym: CD34+CE_2023
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Maria Cristina Mocellin, Maria Cristina Mocellin, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: CD34+CE_2023
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Optimize PBSC Harvest Through Automated Buffy Coat
MeSH Terms: interventions — Blood Component Removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients are defined as subjects affected by a hematological or non-hematological disease for which an autologous stem cells transplantation is recommended. These cases are referred as autologous use of stem cells.
  Interventions: Other: apheresis procedure
- Stem cells donors: Stem cells donors are volunteer healthy subjects who have decided to undergo the procedures needed to collect blood stem cells. These subjects can donate their blood stem cells in favor of a blood relative or, through subscription of a specific registry (IBMDR - International Bone Marrow Donor Registry), to an unknown subject. These cases are referred as allogenic use of stem cells.
  Interventions: Other: apheresis procedure

INTERVENTIONS:
Other: apheresis procedure — collection of hematopoietic stem cells carried out using the single-chamber and continuous mononuclear cell (cMNC) collection system with Spectra Optia (Terumo BCT)

SUMMARY:
All procedures performed during the study will comply with current clinical practice, international and national guidelines. Main object of the study is the PBSC apheresis procedure performed by using the continuous mononuclear cells collection (cMNC) system with Spectra Optia (Terumo BCT), specifically the biological and clinical factors affecting the procedure efficiency.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT), either autologous or allogenic, is a treatment strategy widely used in the onco-hematology field and less often for other diseases1. The most employed source of stem cell is peripheral blood stem cell (PBSC) identified as circulating CD34+ cells and collected by leukapheresis (LP) following mobilization process using granulocyte-colony stimulating factor (G-CSF) alone or in association with chemotherapy and/or plerixafor, the latter in case of poor-mobilizer patients.

The PBSC harvest needs dedicated platform for being properly performed: in our institution the Spectra Optia apheresis system (Terumo BCT) is routinely employed with a continuous mononuclear cells collection (cMNC) system. Spectra Optia (Terumo BCT) is designed to optimize PBSC harvest through automated buffy coat interface identification and management, low volume tubing set, low extracorporeal volumes and support of cMNC processing system3. In the dual-step mononuclear cells collection (MNC) system an intermediate chamber is used to collect white blood cells while returning the majority of platelets to the subject. Then optical sensors detect red blood cells (RBC) overflow and leucocytes are intermittently flushed in the collection bag. The cMNC system differs from the former dual-step system by eliminating the intermediate collection chamber used and thus allowing continuous collection of leucocytes from the buffy coat. This approach appears to be less time consuming, more manageable, and more efficient in returning platelet and RBC to the subject4.

One of the main benchmarks of LP quality is the collection efficiency (CE) defined as the ratio between total CD34+ cells yield in apheresis and total CD34+ cells in the processed blood volume (PBV).

Obtaining the highest possible CE for every LP procedure is critical as long as several studies have shown the importance of targeted CD34+ cells yield in order to assure a safe and rapid haematological recovery after the high dose chemotherapy regimens used in HSCT6. Therefore the objective is to reach the target PBSC yield in the safest and quickest way possible: an high CE allows to reduce the PBV and the procedure length.

The CE values are affected by different factors among which blood sample's physical properties. Such factors have been widely studied in MNC protocol7, but less studies concern the cMNC protocol8. In 147 consecutive apheresis procedures performed both on patients and healthy donors with Spectra Optia (Terumo BCT) with cMNC system, Kondo et colleagues found a moderate positive correlation between CD34+ CE and hematocrit (Ht) and only a very week correlation with white blood cells (WBC) and platelet counts. We would like to confirm these data in a setting of subjects with a predominance of patients over healthy donors, thus evaluating the influence of clinical and biochemical factors on CE for autologous and allogenic hematopoietic stem cell production. Finally we would like to assess a possible pre-LP Ht threshold associated with a sufficient (> 60%) CD34+ CE.

ELIGIBILITY:
Inclusion Criteria:

* Patients and stem cell donors who have been evaluated as suitable for PBSC apheresis and collection, either for autologous or allogenic use
* Patients and stem cell donors that have completed at least one CD34+ apheresis procedure at Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico in Milan.
* Age ≥16 years

Exclusion Criteria:

* Patients affected by Acute Lymphoblastic Leukemia

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will consider consecutive patients and donors referred to the Apheresis Unit within the Transfusional Medicine Department of Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico in Milan (from 1/1/2021 to 31/12/2022) for PBSC collection. Total study population: 113 subjects of which 74 hematological/non hematological patients and 39 stem cell donors.
  Patients are defined as subjects affected by a hematological or non-hematological disease for which an autologous stem cells transplantation is recommended. These cases are referred as autologous use of stem cells.
  Stem cells donors are volunteer healthy subjects who have decided to undergo the procedures needed to collect blood stem cells. These subjects can donate their blood stem cells in favor of a blood relative or, through subscription of a specific registry (IBMDR - International Bone Marrow Donor Registry), to an unknown subject. These cases are referred as allogenic use of stem cells.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
measured by statistical correlation | September 2023 - December 2023
  Impact, measured by statistical correlation, of clinical (age, sex, type of donor, diagnosis, recent RBC transfusion) and biochemical (pre-LP values of Ht, Hb, WBC and PLT) variables on CD34+ CE.
Correlation of clinical | September 2023 - December 2023
  * Correlation of clinical (age, sex, type of donor, diagnosis, recent RBC transfusion) and biochemical variables (pre-LP values of Ht, Hb, WBC and PLT) with an adequate (≥60%) CD34+ CE.
  * Correlation of pre-LP Ht levels and recent (≤ 60 days) RBC transfusion with CD34+ CE, especially in the autologous setting.
  * AUROC (Area Under the ROC Curve) of a pre-LP model based on clinical parameters aimed at predicting an adequate (≥60%) CD34+ CE.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT06308133/Prot_SAP_000.pdf